CLINICAL TRIAL: NCT06551870
Title: Xbox Kinect Sports Versus Nintendo Switch Sports and Their Effects on Body Composition and Physical Performance in Older Female: A Randomized Controlled Trial
Brief Title: Xbox Kinect Sports Versus Nintendo Switch Sports
Acronym: Xb&Nin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Pablo Valdés-Badilla, Researcher, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29/2022
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Healthy People Programs
MeSH Terms: interventions — Exercise; Physical Fitness

STUDY DESIGN:
Intervention Model Description: The study includes an experimental design (randomized controlled trial), double-blind, with repeated measures, parallel groups and a quantitative approach.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Xbox Kinect Sports) (Experimental): The programs were then designed for a duration of 12 weeks (36 sessions), with a 10-minute warm-up consisting of low-intensity aerobic activities and joint mobility, a 40-minute main part and a 10-minute cool-down with static flexibility exercises. The main part of the training sessions included active exergames of volleyball, bowling, boxing, and table tennis, each lasting 8 minutes, with 2 minutes of rest between games. In these active exergames, playing the games will require standing in front of a sensor on a camera under the TV screen in a 3.5-meter-wide range of motion (Li et al., 2021; Marotta et al., 2022).
  Interventions: Other: Physical activity
- Experimental group 2 (Nintendo Switch Sports) (Experimental): The programs were then designed for a duration of 12 weeks (36 sessions), with a 10-minute warm-up consisting of low-intensity aerobic activities and joint mobility, a 40-minute main part and a 10-minute cool-down with static flexibility exercises. In Nintendo Switch Sports in order to run the games of these active exergames you will have to have a controller in your hand that has no cable because it connects via Bluetooth to the console, as in Xbox Kinect Sports you have to play in front of the TV screen (Ramolete et al., 2020). In Nintendo Switch Sports, there will be active exergames of volleyball, bowling, fencing and tennis in the main part, each of 8 min duration, with 2 minutes of rest between games.
  Interventions: Other: Physical activity
- Control group (No Intervention): The control group, the individuals will participate in the assessments (initial and final) and only played board games twice a week for 60 minutes.

INTERVENTIONS:
Other: Physical activity — The complexity of the games will increase as the levels of the sports games advance, which leads to faster movements with greater demands to progress in the sequence of the games, which allows reaching increases in intensity.
  Other Names: Physical fitness
  Arms: Experimental group 1 (Xbox Kinect Sports); Experimental group 2 (Nintendo Switch Sports)

SUMMARY:
The aim of this study will be to compare the effects of Xbox Kinect Sports (XKS) with respect to Nintendo Switch Sports (NSS) and the inactive control group (CG) on body composition (percent body fat and fat-free mass) and physical performance (hand grip strength, HGS; 30 seconds standing in a chair, timed get up and walk, TUG; sit and reach and 2-minute step test) in physically inactive older women. This study will be randomized controlled trial with three parallel groups: XKS (n= 13), NSS (n= 14) and CG (n= 16).

DETAILED DESCRIPTION:
A sealed envelope lottery will be conducted for randomization with a three-arm randomized controlled trial design (XKS, NSS, and CG) with a simple double-blind design (raters and participants). The randomizer's website (https://www.randomizer.org) will be used to carry out the randomization process. The CONSORT guidelines method will be used (Turner et al., 2012). Fifty-two older women initially participated in the intervention. Following previous studies (Hernandez Martínez et al., 2022; Queiroz et al., 2017), the minimum difference needed for significant clinical relevance was a mean difference of 0.60 seconds in TUG, with a standard deviation of 0.20 seconds. An alpha level of 0.05, a power of 85% and an anticipated loss of 20% were considered. The Gpower program (version 3.1.9.6, Franz Faul, Universiät Kiel, Kiel, Germany) was used to calculate the statistical power. The inclusion criteria are as follows: (i) older women, between 60 and 65 years of age; (ii) who did not present cognitive impairment with a score on the Mini-Mental State Examination ≤21 points (Ministerio de Salud, 2013); (iii) who did not present visual difficulty and/or vestibular impairment that would make it difficult to play the games in front of the screen; (iv) who were independent, defined by having at least a score of 43 points on the Chilean Ministry of Health's Preventive Medicine Examination for Older Adults (Ministerio de Salud, 2013); (v) who could meet the attendance requirement of at least 85% of the sessions scheduled for the intervention; (vi) physically inactive who did not meet the international recommendations for moderate (<150 to 300 minutes) or vigorous (<75 to 150 minutes) physical activity (Bull et al., 2020); and (vii) physical condition compatible with the practice of physical activity. As for exclusion criteria, the following were taken into account (i) being afflicted with a disability; (ii) suffering from a musculoskeletal injury or receiving physical rehabilitation therapy, which prevents them from performing their usual physical activity; and (iii) being temporarily or permanently unable to perform physical activity.

By approving the use of the data for scientific purposes by signing an informed consent form, all participants acknowledged the inclusion criteria for the use and treatment of the data. The protocol was created by the Declaration of Helsinki and approved by the scientific ethics committee of the Universidad Católica del Maule, Chile (Approval number: N°29-2022).

ELIGIBILITY:
Inclusion Criteria:

* Older female aged between 60 and 75 years old.
* Presenting the ability to understand and execute direct commands in a contextualized manner.
* Independent, that is, have a score equal to or greater than 43 points in the Preventive Medicine Exam for the Older People (in Spanish, EMPAM) of the Ministry of Health (Ministerio de Salud, 2013).
* Did not present any visual difficulty and/or any vestibular alteration that would hinder the performance of the games in front of the screen-
* Complying with at least 85% attendance at the sessions scheduled for interventions.

Exclusion Criteria:

* Having any disabling disease.
* Those female who have musculoskeletal injuries or who are undergoing physical rehabilitation treatment that prevents their normal physical performance.
* Those who have permanent or temporary contraindications to perform physical activity.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Change from Fat-free mass at 12 weeks | 2 weeks
  This variable is obtained by body composition (bioimpedance), using eight-electrode tetrapolar bioimpedance (InBody 570®, Body Composition Analyzers, South Korea). For each measurement, the guidelines of the International Society for Advances in Kinanthropometry will be followed (Marfell-Jones et al., 2012).
Change from Body fat percentage at 12 weeks | 2 weeks
  This variable will be obtained by body composition (bioimpedance), using eight-electrode tetrapolar bioimpedance (InBody 570®, Body Composition Analyzers, South Korea). For each measurement, the guidelines of the International Society for Advances in Kinanthropometry will be followed (Marfell-Jones et al., 2012).
Change from Maximal isometric handgrip strength at 12 weeks | 2 weeks
  Previous recommendations indicate that maximal isometric handgrip strength (Lupton-Smith et al., 2022), was employed. The best position for testing was found to be sedentary, with the wrist and forearm in a neutral position, the elbow flexed at a 90-degree angle to the side of the body, the spine aligned, and the shoulder in a neutral position. A portable dynamometer (Jamar®, PLUS+, Sammons Preston, Patterson Medical, Warrenville, IL, USA) was used for testing. The dynamometer was placed in the first position, which promotes contact between the first phalanx of the thumb and index finger, to allow a firm grip on the device while preserving proper closure of the metacarpal, palatine, and interphalangeal joints based on hand size. Each participant performed three attempts with each hand after a 120-second rest.
Change from 30-second chair stand test at 12 weeks | 2 weeks
  The 30-second chair stand test (Bruun et al., 2019), which measures the number of repetitions performed standing and sitting in a chair with arms resting on the chest for 30 seconds, will be used to assess lower limb muscle strength and the ability to perform activities of daily living (Jones et al., 1999). The best of the three efforts will be taken into account for the analysis after three attempts, with a recovery of 120 seconds between them.
Change from Timed up-and-go test at 12 weeks | 2 weeks
  The tiemd up-and- go test will be performed according to previous recommendations (Christopher et al., 2021). The individual will be asked to get out of a chair with arm rests, walk down a 3-meter hallway, turn around, and return to the chair. The timed up-and-go is a measure of functional mobility and dynamic balance (Podsiadlo & Richardson, 1991). They are asked to perform three trials and quickly record the best one. Using single-beam photocells (Brower Timing System, Draper, UT, USA), two evaluators will record the time; a statistical analysis of the three best trials will be performed.
Change from Sit-and-reach test at 12 weeks | 2 weeks
  Using the sit-and-reach test, flexibility was assessed (Rikli & Jones, 2013). Subjects sat forward in a chair with a fixed back, one leg bent on the floor and the other left leg straight. Either the left or right leg could be used for comfortable running; however, the post-test measured the same leg as the pre-test. After correcting one position once again, the other bent leg case was assessed for flexibility by running two trials using the highest number to determine the outcome (Lemmink et al., 2003).
Change from 2-minute step test at 12 weeks | 2 weeks
  Cardiorespiratory fitness was measured using the 2-minute step test (Rikli & Jones, 2013). Participants were asked to stand up straight and the average distance between the kneecap and the pelvic bones was marked on a wall with colored tape. Participants performed steps so that their knees were raised above the marked point and the number of repetitions in 2 minutes was recorded (Rikli & Jones, 2013).

SECONDARY OUTCOMES:
Age | 1 week
  In years, through an interview and identity card.
Academic level | 1 week
  Primary, secondary, bachelor, master, PhD. Consulting their curriculum background
Civil status | 1 week
  Married, separated, widow, single, others. Through an interview

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Valdés-Badilla, PhD, Principal Investigator — Universidad Católica del Maule
Locations (1):
- Community center, Osorno, Los Lagos Region, Chile

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared. We will only disseminate the results of the study through scientific papers and presentations at scientific congresses.

REFERENCES:
- [Result] Bruun IH, Mogensen CB, Norgaard B, Schiottz-Christensen B, Maribo T. Validity and Responsiveness to Change of the 30-Second Chair-Stand Test in Older Adults Admitted to an Emergency Department. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):265-274. doi: 10.1519/JPT.0000000000000166. PMID 29227412
- [Result] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Result] Christopher A, Kraft E, Olenick H, Kiesling R, Doty A. The reliability and validity of the Timed Up and Go as a clinical tool in individuals with and without disabilities across a lifespan: a systematic review. Disabil Rehabil. 2021 Jun;43(13):1799-1813. doi: 10.1080/09638288.2019.1682066. Epub 2019 Oct 26. PMID 31656104
- [Result] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Result] Hernandez Martínez, J., Ramirez Campillo, R., Álvarez, C., Valdés Badilla, P. A., Moran, J., & Izquierdo, M. (2022). Effects of active exergames training on physical functional performance in older females. Cultura_Ciencia_Deporte [CCD], 51(17).
- [Result] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Result] Lemmink KA, Kemper HC, de Greef MH, Rispens P, Stevens M. The validity of the sit-and-reach test and the modified sit-and-reach test in middle-aged to older men and women. Res Q Exerc Sport. 2003 Sep;74(3):331-6. doi: 10.1080/02701367.2003.10609099. No abstract available. PMID 14510299
- [Result] Li J, Li L, Huo P, Ma C, Wang L, Theng YL. Wii or Kinect? A Pilot Study of the Exergame Effects on Older Adults' Physical Fitness and Psychological Perception. Int J Environ Res Public Health. 2021 Dec 8;18(24):12939. doi: 10.3390/ijerph182412939. PMID 34948547
- [Result] Lupton-Smith A, Fourie K, Mazinyo A, Mokone M, Nxaba S, Morrow B. Measurement of hand grip strength: A cross-sectional study of two dynamometry devices. S Afr J Physiother. 2022 Sep 26;78(1):1768. doi: 10.4102/sajp.v78i1.1768. eCollection 2022. PMID 36262213
- [Result] Marfell-Jones, M., Olds, T., & De Ridder, J. (2012). International Standards for Anthropometric Assessment (Vol. 137).
- [Result] Marotta N, Demeco A, Indino A, de Scorpio G, Moggio L, Ammendolia A. Nintendo WiiTM versus Xbox KinectTM for functional locomotion in people with Parkinson's disease: a systematic review and network meta-analysis. Disabil Rehabil. 2022 Feb;44(3):331-336. doi: 10.1080/09638288.2020.1768301. Epub 2020 Jun 1. PMID 32478581
- [Result] Ministerio de Salud. (2013). Manual de Aplicación del Examen de Medicina Preventiva del Adulto Mayor. . https://www.minsal.cl/portal/url/item/ab1f81f43ef0c2a6e04001011e011907.pdf
- [Result] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Result] Queiroz, B. M. d., Borgatto, A. F., Barbosa, A. R., & Guimarães, A. V. (2017). Exergame vs. Aerobic Exercise and Functional Fitness of Older Adults: A Randomized Controlled Trial. Journal of physical education and sport, 17, 740.
- [Result] Ramolete, G., Almirante, J., Mondragon, J., Ting, C., Cohen, M., & Custodio, B. (2020). Physical Design Assessment of the Nintendo Switch Controller Configurations. In (pp. 198-205). https://doi.org/10.1007/978-3-030-51038-1_29
- [Result] Richardson, J. T. E. (2011). Eta squared and partial eta squared as measures of effect size in educational research. Educational Research Review, 6(2), 135-147. https://doi.org/https://doi.org/10.1016/j.edurev.2010.12.001
- [Result] Rikli, R. E., & Jones, C. J. (2013). Senior fitness test manual. Human kinetics.
- [Result] Rytterstrom P, Stromberg A, Jaarsma T, Klompstra L. Exergaming to Increase Physical Activity in Older Adults: Feasibility and Practical Implications. Curr Heart Fail Rep. 2024 Aug;21(4):439-459. doi: 10.1007/s11897-024-00675-9. Epub 2024 Jul 18. PMID 39023808
- [Result] Turner L, Shamseer L, Altman DG, Weeks L, Peters J, Kober T, Dias S, Schulz KF, Plint AC, Moher D. Consolidated standards of reporting trials (CONSORT) and the completeness of reporting of randomised controlled trials (RCTs) published in medical journals. Cochrane Database Syst Rev. 2012 Nov 14;11(11):MR000030. doi: 10.1002/14651858.MR000030.pub2. PMID 23152285